CLINICAL TRIAL: NCT03748433
Title: Assessment of the Impact of Real-Time Continuous Glucose Monitoring on People Presenting With Severe Hypoglycaemia
Acronym: AIR-CGM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated early after the interim analysis. It was deemed unethical to offer self-monitored blood glucose to this high risk population
Sponsor: Imperial College London (Other)
Collaborators: London Ambulance Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18HH4609
Record Dates: First submitted 2018-11-07; First posted 2018-11-20 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1; Hypoglycemia Unawareness; Hypoglycemia
Keywords: Real time continuous glucose monitoring; continuous subcutaneous insulin infusion; self monitoring blood glucose; sensor augmented pump; severe hypoglycaemia; hypounaware
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Randomised open-label parallel group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Continuous Glucose Monitoring (CGM) (Experimental): The RT CGM group will receive a Dexcom G6 transmitter and sensors, as well as a structured education refresher focusing on hypoglycaemia avoidance, recognition, and management.
  Interventions: Device: Dexcom G6 CGM
- Self Monitoring Blood Glucose (SMBG) (No Intervention): The SMBG group will additionally undergo blinded CGM at weeks 1 and 2, weeks 4 to 6 and weeks 9 to 12 using the Dexcom G6 system. Participants in this group will be shown how to insert the Dexcom G6 at the first clinic visit and sensors provided so they can do this at home.
- Continuous Subcutaneous Insulin Infusion (CSII) (Experimental): All participants will be re-consented with the choice to continue using RT-CGM for a further 16 weeks or be re-randomised to either receive the Tandem t:slim X2 insulin pump or RT-CGM. Participants randomised to the Tandem t:slim X2 group will be proficiently trained to safely use the Tandem t:slim X2 insulin pump. All participants (Tandem t:slim X2 and RT-CGM) will be provided with Dexcom G6 real time CGM transmitters and sensors for the 16-week second extension phase.
  Interventions: Device: Dexcom G6 CGM; Device: Tandem t:slim X2 Insulin Pump

INTERVENTIONS:
Device: Dexcom G6 CGM — Commercially available Dexcom G6 Continuous Glucose Monitoring
  Arms: Continuous Glucose Monitoring (CGM); Continuous Subcutaneous Insulin Infusion (CSII)
Device: Tandem t:slim X2 Insulin Pump — sensor augmented insulin pump with predictive low glucose suspend
  Arms: Continuous Subcutaneous Insulin Infusion (CSII)

SUMMARY:
This study aims to assess the impact of real-time continuous glucose monitoring on the frequency, duration, awareness and severity of hypoglycaemia in people with type 1 diabetes and a recent history of severe hypoglycaemia, compared to usual care.

DETAILED DESCRIPTION:
Type 1 diabetes (T1DM), which affects 300,000 in the UK, is characterised by autoimmune destruction of the pancreatic beta cells, leading to absolute deficiency of insulin. Management of T1DM requires exogenous insulin administration, aiming for glucose concentrations as close to physiological values as possible. Intensive management of T1DM improves glucose control and reduces the risk of microvascular diabetes complications and cardiovascular disease1. In the UK diabetes consumes more than 10% of the National Health Service budget 2 and in the USA a relatively greater amount is spent on type 1 compared with type 2 diabetes (8.6% of the diabetes budget compared with 5.6% of diabetes prevalence)3. Medication and insulin pump therapy accounts for less than 10% of diabetes expenditure with the majority of costs incurred in the treatment of complications4.

Optimal control remains challenging to achieve and intensive insulin treatment increases the risk of severe hypoglycaemia, with lower glucose values also associated with an increased frequency and severity of moderate hypoglycaemia5, 6. Severe hypoglycaemia is defined as any episode of hypoglycaemia requiring the assistance of a third party actively to treat. Hypoglycaemia is associated with morbidity and even mortality, and places a financial burden on health systems.

Severe hypoglycaemia costs £13million per year in NHS costs7. Between 4 and 10% of deaths in people with type 1 diabetes are attributed to hypoglycaemia and the risk of severe hypoglycaemia increases 6-fold in people with impaired awareness of hypoglycaemia. Avoidance of hypoglycaemia is associated with restoration of hypoglycaemia awareness and this may be enabled by the use of continuous glucose monitoring.

In type 1 diabetes real-time continuous glucose monitoring (CGM) improves overall glucose control in all age groups when used continuously, reduces hypoglycaemia in people with an HbA1c <7.0%, and may reduce severe hypoglycaemia8-10.

The predictive Low-Glucose suspend (PLGS) feature in sensor augmented insulin pumps (SAP) automatically reduces insulin delivery when trends in CGM glucose concentrations predict future hypoglycaemia, and significantly reduces hypoglycaemia without rebound hyperglycaemia compared to SAP without PLGS11.

In England continuous glucose monitoring is supported by NICE for people with type 1 diabetes who are willing to commit to using it at least 70% of the time and to calibrate it as needed, and who have any of the following despite optimised use of insulin therapy and conventional blood glucose monitoring12:

* More than 1 episode a year of severe hypoglycaemia with no obvious preventable precipitating cause.
* Complete loss of awareness of hypoglycaemia.
* Frequent (more than 2 episodes a week) asymptomatic hypoglycaemia that is causing problems with daily activities.
* Extreme fear of hypoglycaemia.
* Hyperglycaemia (HbA1c level of 75 mmol/mol [9%] or higher) that persists despite testing at least 10 times a day

Addressing severe hypoglycaemia, reducing the risk of further episodes and acting promptly to optimise hypoglycaemia awareness are critical in people at high risk.

Continuous subcutaneous insulin pump therapy is supported for adults and children over 12 with type 1 diabetes in whom attempts to achieve target haemoglobin A1c (HbA1c) with multiple daily injections (MDI) have resulted in disabling hypoglycaemia or HbA1c levels have remained high (8.5% [69 mmol/mol] or above) despite high level care12.

ELIGIBILITY:
PRE-REGISTRATION EVALUATIONS

* Episode of severe hypoglycaemia
* Age >18 years
* Diagnosis of type 1 diabetes

INCLUSION CRITERIA

* Adults over 18 years of age
* Severe hypoglycaemia requiring ambulance call-out or emergency department attendance within 2 weeks
* Type 1 diabetes confirmed on the basis of clinical features
* Type 1 diabetes for greater than 3 years

EXCLUSION CRITERIA

* Use of CGM within the last 6 months (except short periods of diagnostic blinded use under clinic supervision). Prior use of Abbott FreeStyle Libre Device is permitted.
* Use of pre-mixed insulin
* No access to smartphone or computer
* Pregnant or planning pregnancy
* Breastfeeding
* Have active malignancy or under investigation for malignancy
* Severe visual impairment
* Reduced manual dexterity
* Unable to participate due to other factors, as assessed by the Chief Investigators

WITHDRAWAL CRITERIA

Participants will be withdrawn if their ability to give informed consent is impaired. Participants will also be withdrawn, at the chief investigators discretion, if glucose control is negatively impacted by the use of either intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Oliver, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Avari P, Ramli R, Reddy M, Oliver N, Fothergill R. Rationale and protocol for the Assessment of Impact of Real-time Continuous Glucose Monitoring on people presenting with severe Hypoglycaemia (AIR-CGM) study. BMC Endocr Disord. 2019 Oct 26;19(1):110. doi: 10.1186/s12902-019-0439-3. PMID 31655586
- See also: NICE Guidelines — https://www.nice.org.uk/guidance/ng17/resources/type-1-diabetes-in-adults-diagnosis-and-management-pdf-1837276469701

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was undertaken in collaboration with the London Ambulance Service. Participants were identified following an episode of severe hypoglycaemia. Following any questions, London Ambulance Services and Emergency Departments obtained verbal consent to share details with study investigators, and sent details to principal investigator through a secure website (NHS.net account). Prrticipants had to be enrolled within two weeks of the severehypoglycaemia episode.
Pre-assignment Details: Once participants were enrolled they were randomised to either real-time CGM (intervention) or self-monitoring of blood glucose (standard care) for 12 weeks.
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring (CGM) | Self Monitoring Blood Glucose (SMBG)
Started | 17 | 18
Completed | 16 | 14
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Population: Baseline demographics are based on the n=30 that completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Glucose Monitoring (CGM) | Self Monitoring Blood Glucose (SMBG) | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38.5 [31.3 to 52.3] | 45.5 [35.3 to 57.8] | 41 [34.3 to 54.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 16 | 14 | 30
Region of Enrollment [Number; unit: participants]
  United Kingdom | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Time Spent in Hypoglycaemia
Description: Percentage time spent in hypoglycaemia (<3.0mmol/L, 55mg/dL)
Time Frame: 12 weeks
Population: Participants who had sufficient data were included in analysis of primary outcome
Measure: Median (Inter-Quartile Range); unit: percentage time
Arm/Group | Continuous Glucose Monitoring (CGM) | Self Monitoring Blood Glucose (SMBG)
Number analyzed (Participants) | 15 | 8
percentage time | 1.8 [0.3 to 3.4] | 3.3 [1.9 to 5.7]

ADVERSE EVENTS:
Time Frame: 1 year Each participant was in the study intervention/control for 3 months
Arm/Group | Continuous Glucose Monitoring (CGM) | Self Monitoring Blood Glucose (SMBG)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 4/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Glucose Monitoring (CGM) (N=16) | Self Monitoring Blood Glucose (SMBG) (N=14)
Unrelated to intervention (Endocrine disorders) | 0 (0) | 4 (4)

LIMITATIONS AND CAVEATS:
The study was terminated early after the interim analysis. It was deemed unethical to offer SMBG to this high risk population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT03748433/Prot_SAP_000.pdf